CLINICAL TRIAL: NCT05457686
Title: The Efficacy of Kinesiology Taping After Total Knee Arthroplasty Surgery
Brief Title: The Efficacy of Kinesiotaping on Pain, Edema and Functionality After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Fevzi Cakmak, assistant proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-08/87
Record Dates: First submitted 2022-07-03; First posted 2022-07-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Knee Arthroplasty; Pain; Edema
Keywords: knee arthroplasty; kinesiotaping
MeSH Terms: conditions — Pain; Edema | interventions — Athletic Tape; Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was designed as blinded, randomized and controlled.the person who evaluates the patients before and after the treatment is blind.In other words,the person evaluating the patients and the person giving the treatment are different.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kinesiology group (Experimental): In the group receiving kinesiology treatment, kinesiotaping is applied to the sub-knee region in accordance with the lymphatic correction technique from the first postoperative day to reduce edema and pain. Accordingly, the proximal part of the tape is placed close to the lymph node. In our study, as stated in the literature, the proximal part of the tape will be adhered to the fibular head area next to the lymph nodes without applying any stretching. Then 5-10% stretching is applied and the distal part is adhered. 2 separate bands are applied so that the strips cross each other (from the medial and lateral of the knee). On the first postoperative day, on the third day, the patients will be taped with kinesio tape and discharged on the fourth day. After discharge, they will be asked to remove the tapes after 3 days as they were taught.
  Interventions: Other: kinesio tape; Other: Exercise
- sham taping group (Sham Comparator): Sham application will be taped with a plaster from the same area on the same days as the kinesio application. No tension will be applied while taping. The difference of the plaster from the kinesiotape is that it does not contain tension and does not allow stretching.
  Interventions: Other: Sham taping; Other: Exercise
- only physical therapy group(control group) (Other): Conservative will be explained on the second day after the operation. Go for a visit with a local cold application 20 times once a day. Ankle pumping exercises, deep breathing exercises, isometric and hip exercises will be planned with a load that can be applied to students who are being applied for bed training.
  Increased the number and allowance of exercises; isotonic knee and exercises that make you feel It will be added. You will be discharged on the 4th day after the surgery on the 2nd or 3rd day. You will do home exercises after discharge. On the 10th day, you will be called for control.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: kinesio tape — According to this, the proximal part of the band is located close to the lymph node. In our study, as stated in the literature, the proximal part of the tape will be adhered to the fibular head area next to the lymph nodes without applying any stretching. Then 5-10% stretching is applied and the distal part is adhered. 2 separate tapes are applied so that the strips cross each other
  Arms: kinesiology group
Other: Sham taping — In the same procedure and time as kinesiotaping, inelastic tape will be used instead of kinesiotape.
  Arms: sham taping group
Other: Exercise — Routine exercise and physiotherapy program applied after knee arthroplasty surgery will be applied

SUMMARY:
In this prospective, randomized controlled trial; To evaluate the effect of kinesiology taping applied for edema on pain, edema and functions in the early period after total knee replacement.Patients who underwent total knee replacement will be included in the 10-day follow-up study.Patients will be divided into three groups by randomization. A conservative postoperative physiotherapy program, which is routinely applied to all groups, will be applied. Thus, no patient will be left without treatment. The first group will be considered as the control group, which will be given only a conservative physiotherapy program.

In addition to the conservative postoperative physiotherapy program, the 2nd group will be taped without applying tension with a plaster and will be considered as the sham group.

In the third group, in addition to the conservative postoperative physiotherapy program, kinesiotaping for payment will be applied.

DETAILED DESCRIPTION:
Patients will be divided into three groups by randomization. A conservative postoperative physiotherapy program, which is routinely applied to all groups, will be applied. Thus, no patient will be left without treatment. The first group will be considered as the control group, which will be given only a conservative physiotherapy program.

In addition to the conservative postoperative physiotherapy program, the 2nd group will be taped without applying tension with a plaster and will be considered as the sham group.

In the third group, in addition to the conservative postoperative physiotherapy program, kinesiotaping for payment will be applied.

It is planned to prevent bias between the groups by giving standard analgesic treatment to all three groups in the postoperative period. In the postoperative period, Paracetamol 10 mg/ml Infusion 3*1, 100 mg tramadol hydrochloride tablet 2*1 and celecoxib capsule 100 mg 2*1 will be routinely administered until the discharge period.

Conservative postoperative physiotherapy program:

Conservative exercise program will be started on the second day after the surgery. All patients will receive an exercise program combined with a 20-minute local cold application once a day. Ankle pumping exercises, deep breathing exercises, isometric knee and hip circumference strengthening exercises, sitting by the bed, timed walking with a tolerable load on the prosthetic side will be recommended.

The number and frequency of exercises were gradually increased; isotonic knee and hip circumference strengthening exercises It will be added. After the drainage of the surgical wound is removed on the 2nd or 3rd day, the patients will be discharged on the 4th postoperative day. All patients will be informed about the conditions and activities that need attention. Patients who continue their home exercise program after discharge will be called for control on the 10th day.

Kinesio taping: In addition to its use in regional pain syndromes in recent years, KT application has also been reported in the literature after various non-orthopedic surgical procedures . Today, after KT application, which is widely used in orthopedics, especially in arthroscopic interventions, no negative effects have been observed on patients, and positive results have been reported, especially in the early period. The investigators aimed to compare this treatment method, which has been shown to be effective in studies performed after total knee arthroplasty, with SHAM taping and conservative postoperative physiotherapy program control group in a prospective randomized comparison.

Kinesiotaping is applied to the sub-knee region in accordance with the lymphatic correction technique in order to reduce edema and pain from the first postoperative day in the group receiving KT treatment.Accordingly, the proximal part of the tape will be placed close to the lymph node.In our study, as stated in the literature, the proximal part of the tape will be adhered to the fibular head area next to the lymph nodes without applying any stretching.Then 5-10% stretching is applied and the distal part is adhered.

The strips are applied as 2 separate bands crossing each other (from the medial and lateral of the knee).The patients will be taped with kinesio tape on the first day and the third day postoperatively, and they will be discharged on the fourth day.

After discharge, participant will be asked to remove the bands after 3 days as instructed.

SHAM taping: Sham application will be taped with a plaster from the same area on the same days as the kinesio application. No tension will be applied while taping. The difference of the plaster from the kinesiotape is that it does not contain tension and does not allow stretching.

Kinesiotaping application; It will be done by a physical therapist who has a kinesiology taping course certificate.

ELIGIBILITY:
Inclusion Criteria:

1. Performing total knee joint arthroplasty due to stage 4 gonarthrosis
2. Agree to participate in the study
3. Having signed the informed consent form

Exclusion Criteria:

1. Presence of malignancy, infection, rheumatological disease
2. Having a tape allergy
3. Having a diagnosis of lymphedema

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
edema | 1 day before surgery
  thigh, knee and leg diameter measurements to be measured with a tape measure
edema | 1 days after surgery
  thigh, knee and leg diameter measurements to be measured with a tape measure
edema | 3 days after surgery
  thigh, knee and leg diameter measurements to be measured with a tape measure
edema | 10 days after surgery
  thigh, knee and leg diameter measurements to be measured with a tape measure

SECONDARY OUTCOMES:
Pain Intensity | 1 day before surgery
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | 1 day after surgery
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | 3 days after surgery
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.
Pain Intensity | 10 days after surgery
  Evaluation of Pain; Visual analog scale (VAS) was used for pain assessment. VAS is in the form of a 10-point Likert scale. Patients are asked to indicate the level of pain, with 0 points as no pain, 5 points as moderate pain, and 10 points as unbearable pain. Increased scores indicate higher pain level.

OTHER OUTCOMES:
Functionality | 1 day before surgery
  Functional assessment: Knee functional assessment will be made using the Oxford Knee Score. The Oxford Knee Score (OKS) was specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is a patient-reported 12-item scale. Each question is scored between 1-5 points from best to severe disability. Turkish validity and reliability has been established.
Functionality | 1 day after surgery
  Functional assessment: Knee functional assessment will be made using the Oxford Knee Score. The Oxford Knee Score (OKS) was specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is a patient-reported 12-item scale. Each question is scored between 1-5 points from best to severe disability. Turkish validity and reliability has been established.
Functionality | 3 days after surgery
  Functional assessment: Knee functional assessment will be made using the Oxford Knee Score. The Oxford Knee Score (OKS) was specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is a patient-reported 12-item scale. Each question is scored between 1-5 points from best to severe disability. Turkish validity and reliability has been established.
Functionality | 10 days after surgery
  Functional assessment: Knee functional assessment will be made using the Oxford Knee Score. The Oxford Knee Score (OKS) was specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is a patient-reported 12-item scale. Each question is scored between 1-5 points from best to severe disability. Turkish validity and reliability has been established.
Measuring knee Joint Range of Motion | 1 day before surgery
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | 1 daysafter surgery
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | 3 days after surgery
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.
Measuring knee Joint Range of Motion | 10 days after surgery
  Knee joint range of motion (ROM) measurement with goniometer is the most commonly used method that provides objective evaluation and error-free measurement in clinical practice. In our study, knee ROM measurements will be made with a goniometer using the neutral zero method. This method is a painless and non-invasive measurement method.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahievran university, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boguszewski D, Tomaszewska I, Adamczyk JG, Bialoszewski D. Evaluation of effectiveness of kinesiology taping as an adjunct to rehabilitation following anterior cruciate ligament reconstruction. Preliminary report. Ortop Traumatol Rehabil. 2013 Oct 31;15(5):469-78. doi: 10.5604/15093492.1084361. PMID 24431257
- [Background] Jongbloed L, van Twist D, Swart N. Kinesio Taping Improves Pain, Range of Motion, and Proprioception in Older Patients With Knee Osteoarthritis. Am J Phys Med Rehabil. 2016 Jan;95(1):e7. doi: 10.1097/PHM.0000000000000393. No abstract available. PMID 26390398
- [Background] Guney Deniz H, Kinikli G, Onal S, et al THU0727-HPR Comparison of kinesio tape application and manual lymphatic drainage on lower extremity oedema and functions after total knee arthroplasty Annals of the Rheumatic Diseases 2018;77:1791.